CLINICAL TRIAL: NCT02729987
Title: Increasing Engagement With and Effectiveness of an Online CBT Based Stress Management Intervention for Employees Through the Use of an Online Facilitated Bulletin Board: Design of a Pilot Randomized Controlled Trial
Brief Title: Increasing Engagement With Online Stress Management Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sussex (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ER/SC587/1
Record Dates: First submitted 2016-03-18; First posted 2016-04-06 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Emotional Stress
Keywords: online; internet; CBT; Stress; Work; Internet based treatment
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Minimum Support Group (MSG) (Experimental): Intervention group with 8 week access to the online stress management programme with minimal support from a coach (WorkGuru).
  Interventions: Behavioral: WorkGuru
- Discussion Group (Experimental): Intervention group with 8 week access to the online stress management programme with minimal support from a coach, plus access to an online facilitated messaging board (WorkGuru).
  Interventions: Behavioral: WorkGuru
- Waiting List Control (WLC) (No Intervention): Control group with access to the intervention after 16 weeks

INTERVENTIONS:
Behavioral: WorkGuru — A multi-modal stress management intervention accessed over 8 weeks, incorporates CBT, positive psychology and Mindfulness. Delivered via the internet.
  Arms: Discussion Group; Minimum Support Group (MSG)

SUMMARY:
The purpose of this pilot study is to explore the effect of an online facilitated discussion group on engagement with a stress management intervention delivered to employees in the UK via the Internet. The investigators primary hypothesis is that the intervention group with access to an online facilitated discussion group (delivered via a message board) will show greater engagement than the intervention group that does not have access to the discussion group. The investigators also hypothesise that participants in the intervention groups will improve significantly on psychological distress and subjective wellbeing measures compared to the waiting list control group, and that the group with access to the online facilitated discussion group will show the greatest improvement.

DETAILED DESCRIPTION:
The aim of the pilot study is to identify and address some of the challenges of delivering online psychological interventions in the workplace. There is clear research evidence for the delivery of online psychological interventions within clinical settings (e.g. Andersson & Cuijpers, 2009), but this evidence does not translate to online interventions delivered in work settings (e.g. Geraedts, Kleiboer, Twisk, Wiezer, van Mechelen, & Cuijpers, 2014). Evidence suggests that one of the barriers to the efficacy of online interventions may be the low level of engagement and adherence (Cavanagh & Millings, 2013). This study aims to address this by asking the question: "How can we increase engagement with and adherence to an online intervention delivered in the workplace?"

The pilot study is a three-arm RCT comparing a minimal guided online Cognitive Behaviour Therapy (CBT) based stress management intervention (WorkGuru) delivered with and without an online facilitated bulletin board, to a waiting list control. Both active conditions will have access to an online programme with minimal support from a coach. The discussion group condition will also have access to a facilitated online bulletin board. Up to 90 employees from UK based organisations will be recruited to the study.

Inclusion criteria will include age 18 or over, elevated levels of stress (defined as 1SD above the mean norm on the PSS-10 scale), access to a computer or tablet, and the Internet. The primary outcome measure will be engagement, as defined by the number of logins to the site; secondary outcome measures will include further measures of engagement (the number of pages visited, the number of modules completed and self-report engagement) and measures of effectiveness (psychological distress and subjective wellbeing). Possible moderators will include measures of intervention quality (satisfaction, acceptability, credibility, system usability), time pressure, goal conflict, level of distress at baseline, and job autonomy. Measures will be taken at baseline, 2 weeks (credibility and expectancy measures only), 9 weeks (completion of intervention) and 16 weeks (follow-up). Analyses will be conducted on intention to treat and per protocol principles. Data will be collected electronically using Qualtrics survey software.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or over
* Employed by a participating organisation, ≥ 20 on the Perceived Stress Scale
* Access to a computer/table and the internet

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of log-in to the site | 9 weeks
  number of times participants log in to the website

SECONDARY OUTCOMES:
Number of modules completed | 9 weeks
  number of modules completed
Number of pages visited | 9 weeks
  number of pages visited
Self-report engagement | 9 weeks
  1 item self-report engagement
Depressions, anxiety and stress | baseline, 9 weeks and 16 weeks
  Depression, Anxiety and Stress Scale (DASS-21)
Well-being at work | baseline, 9 weeks and 16 weeks
  16-item Institute of Work Psychology Multi Affect Indicator

CONTACTS AND LOCATIONS:
Overall Officials: Stephany Carolan, MSc, Principal Investigator — University of Sussex
Locations (1):
- WorkGuru, Brockenhurst, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Andersson G, Cuijpers P. Internet-based and other computerized psychological treatments for adult depression: a meta-analysis. Cogn Behav Ther. 2009;38(4):196-205. doi: 10.1080/16506070903318960. PMID 20183695
- [Background] Cavanagh, K., & Millings, A. (2013). Increasing engagement with computerised cognitive behavioural therapies. ICST Transactions on Ambient Systems, 13(2), e3. http://doi.org/10.4108/trans.amsys.01-06.2013.e3
- [Background] Geraedts AS, Kleiboer AM, Twisk J, Wiezer NM, van Mechelen W, Cuijpers P. Long-term results of a web-based guided self-help intervention for employees with depressive symptoms: randomized controlled trial. J Med Internet Res. 2014 Jul 9;16(7):e168. doi: 10.2196/jmir.3539. PMID 25008127
- [Derived] Carolan S, Harris PR, Greenwood K, Cavanagh K. Increasing engagement with an occupational digital stress management program through the use of an online facilitated discussion group: Results of a pilot randomised controlled trial. Internet Interv. 2017 Aug 24;10:1-11. doi: 10.1016/j.invent.2017.08.001. eCollection 2017 Dec. PMID 30135747
- [Derived] Carolan S, de Visser RO. Employees' Perspectives on the Facilitators and Barriers to Engaging With Digital Mental Health Interventions in the Workplace: Qualitative Study. JMIR Ment Health. 2018 Jan 19;5(1):e8. doi: 10.2196/mental.9146. PMID 29351900
- [Derived] Carolan S, Harris PR, Greenwood K, Cavanagh K. Increasing engagement with, and effectiveness of, an online CBT-based stress management intervention for employees through the use of an online facilitated bulletin board: study protocol for a pilot randomised controlled trial. Trials. 2016 Dec 15;17(1):598. doi: 10.1186/s13063-016-1733-2. PMID 27978858
- See also: Stress management intervention — http://workguru.org